CLINICAL TRIAL: NCT02127021
Title: Prospective Study for the Effects of High Dose Pancreatic Enzyme Replacement Therapy on Body Weight, Quality of Life, and Nutritional Assessment After Pancreatoduodenectomy
Brief Title: The Effects of High Dose Pancreatic Enzyme Replacement Therapy After Pancreatoduodenectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-1401-145-552
Record Dates: First submitted 2014-04-03; First posted 2014-04-30 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2017-12

CONDITIONS: Pancreaticoduodenectomy
Keywords: Pancreaticoduodenectomy; Nutritional Status; Quality of Life; Biochemical Marker

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Norzyme® 40000 IU (Experimental): Single capsule of Norzyme® 40000 IU will be prescribed three times a day while taking a meal meal.
  Interventions: Drug: Norzyme® 40000 IU
- Placebo (Placebo Comparator): Single capsule of placebo drug with the same appearance of Norzyme® 40000 IU will be prescribed three times a day while taking a meal meal. The formulation and the form of placebo is same with the Norzyme® 40000 IU. Placebo contains microcrystalline cellulose as the main component, titanium oxide, colloidal silica, yellow iron oxide, brown iron oxide, black iron oxide, magnesium stearate, triethyl citrate, talc, and simethicone emulsion in very small amount
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Norzyme® 40000 IU — A kind of pancreatic enzyme supplement containing lipase: 40,000 FIP, amylase: 25,000 FIP, and protease: 1,500 FIP Single capsule of Norzyme® 40000 IU will be prescribed three times a day while taking a meal meal
  Other Names: Norzyme
  Arms: Norzyme® 40000 IU
Drug: Placebo — Single capsule of placebo drug with the same appearance of Norzyme® 40000 IU will be prescribed three times a day while taking a meal meal.
  Arms: Placebo

SUMMARY:
Up to now, the studies concerning nutritional assessment after pancreatic resection were rare. The low-dose pancreatic enzyme treatment after pancreatectomy showed no significant benefit in terms of nutritional status. This study is a multicenter randomized phase IV study by using high-dose Norzyme® (40,000 IU) to evaluate quality of life and nutritional status after pancreaticoduodenectomy.

DETAILED DESCRIPTION:
There are not enough studies evaluating nutritional parameters in patients with pancreatic resection. After pancreatic surgery, there are several ways to improve patient condition in terms of quality of life including nutrition.

In the investigators previous study, pancreatic enzyme supplement through the administration of Norzyme® 25000 IU containing lipase 25000 IU, amylase 22500 IU, and protease 1250 IU after various type of pancreatectomy to improve quality of life and nutritional status failed to prove its effectiveness. After administration of low-dose Norzyme® (25000 IU), some patients showed weight gain, but statistically significant conclusions were not obtained mainly because of various types of pancreatectomy and low supplementary dosage of pancreatic enzyme.

Therefore, the investigators design this study to find out the effect of high-dose Norzyme® (40000 IU) on weight gain, quality of life, stool habit change, and nutritional status in patients with pancreaticoduodenectomy. The investigators will evaluate the effectiveness and adequacy of high-dose pancreatic supplementary treatment through a randomized, placebo-using, single-blinded, and multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* ECOG performance status : 0,1,2
* Patients who underwent pancreaticoduodenectomy or pylorus preserving pancreaticoduodenectomy
* stool elastase ≤200, preoperatively and postoperatively
* Patients consented to this study

Exclusion Criteria:

* Patients with comorbidities such as liver cirrhosis, chronic renal failure, heart failure, and inflammatory bowel disease which can affect the assessment of quality of life or nutritional status
* Patients underwent major abdominal organ surgery such as gastrectomy and colon resection which can affect the assessment of quality of life or nutritional status
* Patients with locoregional recurrence or distant metastasis
* Patients which were not able to progress diet and medication within 10 days after surgery
* Patients with pork allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2014-04; Primary Completion 2017-09-07 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in body weight at 3 months after medication | 3 months after medication
  Body weight will be measured 3 times during the entire study period, once preoperatively and two times postoperatively. After surgery, weight will be measured before medication and at the 3 months after medication.These serial weight measurements will be analyzed to figure out changes in body weight over time.

SECONDARY OUTCOMES:
Change from Baseline in Nutritional Status at 3 months after medication | 3 months after medication
  To assess the nutritional status of the patient underwent pancreaticoduodenectomy by testing fasting blood glucose, C-peptide, Insulin, Hb A1c, serum protein, serum albumin, serum pre-albumin, and transferrin
Change from baseline in stool habit at 3 months after medication | 3 months after medication
  To check change from baseline in stool habit at 3 months after medication

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Jang, M.D., PhD., Study Chair — Seoul National University Hospital; Jin-Young Jang, M.D., PhD., Principal Investigator — Seoul National University Hospital
Locations (6):
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam, Bundang-gu
  - Center for Liver Cancer, National Cancer Center, Goyang-si, Gyeonggi-do
  - Dongguk University Ilsan Medical Center, Goyang, Kyeonggi
  - Department of Surgery, Seoul National University College of Medicine, Seoul
  - Chung-Ang University Hospital, Seoul
  - Kangnam Severance Hospital, Seoul

REFERENCES:
- [Derived] Kim H, Yoon YS, Han Y, Kwon W, Kim SW, Han HS, Yoon DS, Park JS, Park SJ, Han SS, Lee SE, Choi SH, Han IW, Kim E, Jang JY. Effects of Pancreatic Enzyme Replacement Therapy on Body Weight and Nutritional Assessments After Pancreatoduodenectomy in a Randomized Trial. Clin Gastroenterol Hepatol. 2020 Apr;18(4):926-934.e4. doi: 10.1016/j.cgh.2019.08.061. Epub 2019 Sep 12. PMID 31520730